CLINICAL TRIAL: NCT01291927
Title: Comparison of Pancreas-sparing Duodenectomy With Pancreatoduodenectomy for Early-stage Periampullary Carcinoma:A Prospective Non-Randomized Trial
Brief Title: Pancreas-sparing Duodenectomy Versus Pancreatoduodenectomy for Early-stage Periampullary Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Institute of Hepatobiliary Surgery, Southwest Hospital (Ping Bie), Institute of Hepatobiliary Surgery, Southwest Hospital ,Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBS-PSU-001
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-01

CONDITIONS: Periampullary Carcinoma Nos
Keywords: Periampullary carcinoma; Pancreas-sparing Duodenectomy; pancreaticoduodenectomy; lymphadenectomy
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pancreas-sparing duodenectomy (Experimental)
  Interventions: Procedure: Pancreas-sparing duodenectomy
- Pancreaticoduodenectomy (Active Comparator)
  Interventions: Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Pancreas-sparing duodenectomy — Pancreas-sparing duodenectomy for periampullary carcinoma is defined as resection of the descending segment of duodenum; resection of papilla of Vater; reimplantation of bile and pancreatic ducts and reconstruction of duodenum.The Japan Pancreatic Society (JPS) system for numbering of lymph node stations was adopted for accurate description of the surgery and pathological assessment.The standard lymph node groups removed as part of PSD were the anterior pancreatoduodenal groups (JPS LN17), the posterior pancreatoduodenal groups (JPS LN13), the dextroinferior nodes of the hepatoduodenal ligament node groups (JPS LN12), the infrapyloric node (JPS LN6), the nodes around the anterior aspect of the common hepatic artery (JPS LN8) and the nodes on the right side of the SMA (JPS LN14).
  Other Names: PSD
  Arms: Pancreas-sparing duodenectomy
Procedure: Pancreaticoduodenectomy — The surgical technique used for standard PD has been described before. Standard PD included clearance of all soft tissues and lymphatics immediately to the left of the superior mesenteric artery, as well as removal of the lymphoareolar tissue along the proximal hepatic artery.
  Other Names: PD
  Arms: Pancreaticoduodenectomy

SUMMARY:
The purpose of this study is to investigate the feasibility, safety, and long-term prognosis of pancreas-sparing duodenectomy with regional lymphadenectomy in the treatment of early-stage (pTis/pT1/pT2) periampullary carcinoma with or without lymph node metastasis

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is commonly used for periampullary carcinoma (PC). In recent years, morbidity and mortality rates following PD have decreased, but the operative stress induced by pancreatectomy is considerable. Less-invasive surgery should thus be elected for PC without pancreatic and diffuse lymph node involvement. From the perspective of organ-preserving resection, pancreas-sparing duodenectomy (PSD) represents an attractive option for selected periampullary tumors, and offers an alternative to PD.

Previous reports have described PSD for benign, premalignant and some selected malignant conditions of duodenum, and have emphasized this procedure as a safe and effective treatment associated with good quality of life. However, use of PSD for PC is still controversial.Available data about PSD for PC and published data from the follow-up evaluation in the literature are still limited.

Given the fact that 20%-60% pT1/pT2 patients have regional lymph node metastasis, regional lymph node dissection should be essential for PC. However, lymphadenectomy has never been promoted as a regular procedure of PSD.The aim of the present study was to investigate the feasibility, safety, and long-term results of PSD with regional lymphadenectomy for early-stage (pTis/pT1/pT2) periampullary cancers.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven periampullary carcinoma (including cancers of distal common bile duct, ampulla or papilla of Vater)
* Pre- and intra-operative stage(CT, EU stage):pTis or pT1 or pT2, N0 or N1, M0
* ASA score: < 3
* Liver function:Child-Pugh A
* No history of other cancers
* No history of preoperative chemotherapy or radiotherapy
* Written informed consent

Exclusion Criteria:

* There are concurrent cancers or the patients have been treated due to other type of cancers before diagnosed as periampullary carcinoma
* Pre- and intra-operative stage: more advanced than T2,or with remote metastasis
* The Patients received other non-surgical therapy, such as chemotherapy, immunotherapy, radiotherapy or endoscopic therapy
* The Patients received upper abdominal surgery
* ASA score: ≥ 3
* Liver function:Child-Pugh B or C
* Pregnancy patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  It is an average time peroid.

SECONDARY OUTCOMES:
Number of Patients with early postoperative complications as a Measure of Safety and Tolerability | up to 2 weeks
  Early postoperative complications consist of gastrointestinal/abdominal bleeding, pancreatic leakage, encephalopathy, delayed gastric emptying, diabetes mellitus and wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Ping Bie, M.D.,Ph.D., Study Director — Institute of Hepatobiliary Surgery, Southwest Hospital, Third Military Medical University; Geng Chen, M.D.,Ph.D., Principal Investigator — Institute of Hepatobiliary Surgery, Southwest Hospital, Third Military Medical University
Locations (1):
- Institute of Hepatobiliary Surgery, Southwest Hospital,Third Military Medical University, Chongqing, Chongqing Municipality, China